CLINICAL TRIAL: NCT03610321
Title: Lipid-lowering Effects of Gefarnate in Statin-treated Coronary Heart Disease Patients With Residual Hypertriglyceridemia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201867
Record Dates: First submitted 2018-07-26; First posted 2018-08-01 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Gefarnate; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Statin group (Active Comparator): Receiving statin treatment (atorvastatin 20 mg or rosuvastatin 10 mg, once daily, oral) only for 1 month.
  Interventions: Drug: Statin
- Gefarnate group (Experimental): Combined treatment with statins (atorvastatin 20 mg or rosuvastatin 10 mg, once daily, oral) and gefarnate (100 mg, three times daily, oral) for 1 month.
  Interventions: Drug: Gefarnate; Drug: Statin

INTERVENTIONS:
Drug: Gefarnate — Gefarnate (100 mg, three times daily, oral) treatment for 1 month.
  Arms: Gefarnate group
Drug: Statin — Statin treatment (atorvastatin 20 mg or rosuvastatin 10 mg, once daily, oral) for 1 month.

SUMMARY:
Dyslipidemia is an independent risk factor for cardiovascular events. Statins have become the cornerstone for the prevention and treatment of atherosclerotic vascular diseases. However, after the comprehensive control of the traditional risk factors, including unhealthy lifestyle, hypercholesterolemia, hypertension, hyperglycemia and obesity, there is still a high risk of residual cardiovascular disease in patients with dyslipidemia. Triglyceride elevation is the most common type of dyslipidemia and constitutes an important component of cardiovascular residual risk.

The geraniol has a variety of pharmacological effects, such as anti-inflammatory, antioxidant, regulating cell apoptosis. Recent studies have confirmed that geraniol plays an important role in regulating glucose and lipid metabolism, and may have a synergistic role with statins. Gefarnate Tablets is a kind of anti-ulcer and gastritis treatment. It can increase the defense ability of gastric mucosa by improving the prostaglandin level and the concentration of amino hexose in the gastric mucosa. Geraniol is the main components of Gefarnate Tablets. In the previous study, the investigators found that geraniol induced autophagy through the SIRT1-AMPK-mTOR pathway and accelerated the degradation of triglycerides in liver cells, thus reducing the level of triglyceride in the serum of high fat diet mice. 6 patients with hyperlipidemia were received Gefarnate Tablets (100mg/ times, 3 times per day). A month later, the levels of serum triglyceride, total cholesterol, and low density lipoprotein cholesterol were decreased significantly. However, the above results need to be confirmed by the larger clinical research.

Therefore, the aim of this study is to evaluate the effect of Gefarnate Tablets on blood lipid levels in patients with hypertriglyceridemia and coronary heart disease treated with statins, provide more options for the treatment of lipid lowering treatment, reduce the risk of cardiovascular remnant, and improve the long-term prognosis of the coronary heart disease patients with residual hypertriglyceridemia.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease
* Treatment with statins for more than 1 month
* Plasma triglyceride level more than 1.7mmol/L

Exclusion Criteria:

* Atherosclerotic cardiovascular disease (ASCVD) patients with high risk
* Patients with active liver disease or unexplained elevated levels of aminotransferase
* Patients with prostatic hypertrophy or those with prostaglandin drugs such as glaucoma
* Creatinine clearance < 30ml/min
* an allergy to any component of Gefarnate Tablets or statin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Triglyceride change from baseline | 1 month
  Triglyceride change from baseline

SECONDARY OUTCOMES:
Total cholesterol and low density lipoprotein cholesterol changes from baseline | 1 month
  Total cholesterol and low density lipoprotein cholesterol changes from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- the first affiliated hospital of Harbin medical university, Harbin, Heilongjiang, China